CLINICAL TRIAL: NCT07008937
Title: The Effect of Balneotherapy on the Inflammatory Process and Quality of Life in Patients With Knee Osteoarthritis
Brief Title: The Effect of Balneotherapy on Knee Osteoarthritis
Acronym: Balneotherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Figen Tuncay, Clinical Professor, Head of Physical Medicine and Rehabilitation, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-06/63
Record Dates: First submitted 2025-05-23; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Balneology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balneotherapy group (group 1) (Experimental): Group 1 -Patients in the research group will receive geothermal treatment (spa therapy) for 20 minutes daily for 15 days.
  Interventions: Other: Balneotherapy
- Control Group (group 2) (Other): Group 2- Patients in the control group will be followed up with only a home exercise program
  Interventions: Other: home exercise program

INTERVENTIONS:
Other: Balneotherapy — For balneotherapy, patients will be treated in a thermal pool for 15-20 minutes daily, with full-body immersion, for a total of 15 days.
  For control, Volunteers in the control group will only receive a home exercise program. They will be called in for a check-up every five days to confirm that the home program is being followed correctly. In this way, the volunteers in the control group will not be left completely without treatment.
  Arms: Balneotherapy group (group 1)
Other: home exercise program — home exercise program
  Arms: Control Group (group 2)

SUMMARY:
Osteoarthritis (OA) is a chronic degenerative disease characterized by the breakdown and repair processes of the cartilage structure in synovial joints. Balneotherapy is one of the most commonly applied treatment methods in patients with OA. It is used to reduce pain and stiffness, improve joint mobility and quality of life, and prevent disease progression. Hyperthermia caused by balneotherapy activates the sympathetic nervous system and the hypothalamic-pituitary-adrenal (HPA) axis. After heat stress, HSp levels in the blood increase, triggering the HSp-cytokine-HPA-cortisol anti-inflammatory feedback mechanism, resulting in an anti-inflammatory effect and neuroendocrine immune regulation.

In various pathologies associated with low-grade inflammation-especially rheumatic diseases-balneotherapy and mud therapy have been reported to decrease serum concentrations of pro-inflammatory cytokines such as TNF-α and IL-1β. Serum COMP levels are elevated in OA patients. There is evidence that measuring COMP levels could serve as a prognostic marker for the development of OA in patients with chronic knee pain. It is evaluated not only as a cartilage marker but also as an indicator of synovial inflammation.

The aim of this study is to evaluate the response to inflammation and stress in patients with knee OA by examining the levels of CRP, IL-1 beta, COMP, and HSp following balneotherapy treatment. Additionally, changes in patients' quality of life and functional status after balneotherapy will also be evaluated.Fifty patients with primary osteoarthritis who meet the inclusion criteria and are receiving inpatient or outpatient treatment in the Physical Medicine and Rehabilitation clinic will be included in the study. It is planned to include 30 patients in the treatment group and 20 patients in the control group. Pain will be assessed using VAS, physical function and stiffness using WOMAC, and quality of life using the SF-36 scale. To determine the serum levels of COMP, IL-1 beta, CRP, and HSp70, blood samples will be collected under standard conditions from patients in a fasting state between 8:00-9:00 AM. Biochemical markers will be evaluated using ELISA kits.

For balneotherapy, patients will be treated in a thermal pool for 15-20 minutes daily, with full-body immersion, for a total of 15 days.

DETAILED DESCRIPTION:
In various pathologies associated with low-grade inflammation-especially rheumatic diseases-balneotherapy and mud therapy have been reported to decrease serum concentrations of pro-inflammatory cytokines such as TNF-α and IL-1β. COMP (cartilage oligomeric matrix protein) contributes to the stabilization of the collagen network by binding to collagen IX. Serum COMP levels are elevated in OA patients. There is evidence that measuring COMP levels could serve as a prognostic marker for the development of OA in patients with chronic knee pain. In OA, elevated IL-1 levels increase matrix metalloproteinase (MMP) levels and reduce TIMP synthesis. IL-1 plays the major role in the production of destructive enzymes. It also increases the synthesis of PGE2, which promotes inflammation and bone resorption. While severe heat stress causes cellular damage and cell death, the mild heat stress seen in balneotherapy induces a heat shock response. Following stress stimuli such as heat and inflammation, intracellular synthesis of heat shock proteins (HSp) increases, and there is a significant transition to the extracellular space. After heat stress, HSp levels in the blood increase, triggering the HSp-cytokine-HPA-cortisol anti-inflammatory feedback mechanism.

To investigate the effect of balneotherapy on these markers; Male and female patients aged between 50 and 80 years with knee osteoarthritis (KOA) at stages 2 to 4 according to the Kellgren-Lawrence classification (Kellgren and Lawrence, 1957), based on imaging performed within the past year, were included in the study. The study is a parallel-group randomized controlled trial conducted at the Thermal Center of Kırşehir Ahi Evran Training and Research Hospital. The RCT was approved by the Ethics Committee of Kırşehir Ahi Evran University; The study is planned to start in July 2025 and to be completed in November 2025. Participants will be randomly assigned to the intervention and control groups in a 1:1 allocation ratio.

The intervention group is planned to receive therapy 5 days a week, at the same time each morning, for 15-20 minutes per session, totaling 15 sessions. The control group will receive a home exercise program and simple analgesic treatment such as paracetamol. Both control and intervention groups received a booklet with general information and advice about how to improve the symptoms and progression of knee osteoarthritis. Data will be expressed as mean ± SD. Statistical analyses will be performed using SPSS version 22. A p-value of <0.05 will be considered statistically significant. Wilcoxon test will be used for comparisons before and after treatment, and Mann-Whitney U test will be used for comparisons between groups.

ELIGIBILITY:
Inclusion Criteria:

* Being over 50 years old
* Patients diagnosed with knee OA
* At stages 2-to-4 according to the Kellgren- Lawrence classification
* Patients who agree to receive balneotherapy treatment

Exclusion Criteria:

* Neoplasia
* Infections
* Uncompensated cardiac or pulmonary problems
* Total knee arthroplasty
* Inflammatory joint diseases (e.g., RA, AS)
* Intra-articular injections in the past 6 months
* Corticosteroids or anti-cytokine therapy
* Patients with a BMI over 30 kg/m2

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
the serum levels of COMP, IL-1 beta, CRP, and HSp70 | Levels of COMP, IL-1 beta, CRP, and HSp70 will be measured one day before the start of the balneotherapy (baseline) and one day after completing the 15-session therapy (15 days)
  Before starting the treatment and one day after completing the 15-session balneotherapy, levels of COMP, IL-1 beta, CRP, and HSp70 will be measured in the intervention group.

SECONDARY OUTCOMES:
Visual Analogue Scale | Assessments will be made at baseline and at the end of treatment (15 season ) completion (15 days) for both groups.
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Western Ontario ve McMaster Universities Osteoartrit (WOMAC) | Assessments will be made at baseline and at the end of treatment (15 season ) completion (15 days) for both groups.
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Higher scores indicate worse pain, stiffness, and functional limitations.
Short -Form 36 | Assessments will be made at baseline and at the end of treatment (15 season ) completion (15 days) for both groups.
  The SF-36 is used to objective measure of the quality of life.It comprises 36 questions that cover eight domains of health. Higher scores indicate better health status.

IPD SHARING:
Plan to Share IPD: No